CLINICAL TRIAL: NCT06546735
Title: Randomized, Double-blind, Double-masked, Parallel-group, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Two Fixed-dose Combinations in Men with Lower Urinary Tract Symptoms Associated with Benign Prostatic Hyperplasia.
Brief Title: Efficacy and Safety of Two Fixed-dose Combinations in Men with Lower Urinary Tract Symptoms Associated with Benign Prostatic Hyperplasia. (BENIPRO)
Acronym: BENIPRO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF185
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia with Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Test Group: N0728 - each participant should take 2 tablets a day, in the morning, after feeding. In a blinded manner, participants in the test group will be required to take 1 tablet of the test drug (N0728) and 1 tablet of placebo of alpha-adrenergic antagonists.
  Comparator Group: alpha-adrenergic antagonists - Participants in the control group will be required to take 1 tablet of the comparator drug (alpha-adrenergic antagonists) and 1 tablet of the placebo of the test drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N0728 (Experimental): in the test group will be required to take 1 tablet of the test drug (N0728) and 1 tablet of placebo of Vesomni®. 2 tablets a day, in the morning, after feeding for 84 days.
  Interventions: Drug: N0728
- Vesomni® (Active Comparator): in the control group will be required to take 1 tablet of Vesomni® and 1 tablet of the placebo of the test drug. 2 tablets a day, in the morning, after feeding for 84 days.
  Interventions: Drug: Vesomni®

INTERVENTIONS:
Drug: N0728 — 1 tablet of the test drug (N0728) and 1 tablet of placebo of Vesomni®.
  Arms: N0728
Drug: Vesomni® — 1 tablet of the comparator drug Vesomni® and 1 tablet of the placebo of the test drug.
  Arms: Vesomni®

SUMMARY:
The clinical trial to evaluate the fixed-dose combination (N0728), with the aim of providing the Brazilian market with an alternative, potentially effective, safe and convenient therapeutic approach for the treatment of Lower Urinary Tract Symptoms (LUTS) in men with Benign Prostatic Hyperplasia (BPH). The fixed-dose combination has synergistic action between drugs from different classes and offers significant potential advantages, such as better adherence to treatment. The trial will assess the non-inferiority in efficacy and safety of the proposed fixed-dose combination compared to alpha-adrenergic antagonists.

DETAILED DESCRIPTION:
This is a phase 3, prospective, randomized, multicenter, double-blind, double-masked, parallel group clinical trial to evaluate the efficacy and safety of the fixed-dose combination (FDC) of (N0728) in the treatment of men with moderate to severe storage symptoms (urgency, increased urinary frequency, urge urinary incontinence) and emptying symptoms (weak urine stream, straining or hesitation in urination, sensation of incomplete urination, terminal drip), associated with benign prostatic hyperplasia (BPH).

The trial will have a total duration of a maximum of 116 days (approximately 16 weeks): up to 4 weeks of screening and 12 weeks (± 4 days) of treatment. Potential participants will be screened at Visit -1. Participants who are currently using alpha-blockers will be required to undergo a period of 2 weeks of washout, thus ensuring the homogeneity of the population at the entry of the trial. All participants will have up to 2 weeks to perform the planned laboratory and imaging tests. At the randomization visit (RV), if eligible, participants will be randomized in a 1:1 ratio and begin trial treatment in a double-blind manner. During the treatment period, participants will return to the study site for two intermediary visits (Visit 1 and 2), and after completing 12 weeks of treatment participants are expected to return for the Final Visit (FV).

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all purposes of the trial by signing and dating the Informed Consent Form in two copies.
* Men ≥40 years of age.
* History of overactive bladder symptoms (urinary frequency and urgency with or without urinary incontinence) and LUTS for at least 3 months due to BPH.
* History of urinary symptoms (≥1 urgency/24-hour episode and ≥8 urination/24-hour) for at least 3 months prior to screening.

Exclusion Criteria:

* Participant who has received mirabegrone or antimuscarinics for the treatment of LUTS within the last 30 days prior to the Screening Visit.
* Participant with evidence of lower urinary tract infection (UTI), confirmed by a culture >100,000 CFU/mL. Should a participant present with a UTI at screening, they may be screened again after successful UTI treatment (confirmed by negative urine culture).
* Participant with symptomatic UTI, prostatitis, or chronic inflammation (such as interstitial cystitis, bladder stones, prior pelvic radiation therapy, or previous or current malignancy within the boundaries of the pelvis, including bladder, prostate, and rectum).
* History of recurrent UTI (2 episodes in the last 6 months or 3 episodes in the last year).
* Participant who has neurogenic bladder (spinal cord injury, multiple sclerosis, Parkinson's, etc.).
* Participant with a previous diagnosis of diabetic neuropathy.
* History of previous open, robotic, or minimally invasive prostate surgery (including transurethral procedures), or reconstructive bladder surgery.
* Participant with planned pelvic or prostate surgery during the trial period.
* Participant with planned cataract or glaucoma surgery during the trial period.
* Participant with significant stress incontinence or post-surgical prostate incontinence as determined by the Investigator.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2026-11-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
The mean number of urgency episodes per day | 12 weeks
  Change from baseline (RV) to the end of 12 weeks of treatment (FV) in the mean number of urgency episodes per day, based on the 3-day voiding diary.

SECONDARY OUTCOMES:
The mean number of voids per day | 12 weeks
  Change from baseline (RV) to the end of 12 weeks of treatment (FV) in the mean number of voids per day, based on the 3-day voiding diary.
The mean number of incontinence episodes per day | 12 weeks
  Change from baseline (RV) to the end of 12 weeks of treatment (FV) in the mean number of incontinence episodes per day, based on the 3-day voiding diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No